CLINICAL TRIAL: NCT05966051
Title: MuLtidimensional School-based and Family Involved interVentions, to Promote a hEalthy and Sustainable LifestYle for the Childhood Obesity Primary Prevention: the LIVELY Study
Brief Title: MuLtidimensional School-based and Family interVentions to Promote hEalthy and Sustainable LifestYle for the Childhood
Acronym: LIVELY
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: IRFMN-8979; F13C22001210007 (Other: University of Pavia)
Record Dates: First submitted 2023-03-23; First posted 2023-07-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Childhood Obesity
Keywords: Childhood Obesity Prevention; Childhood Obesity determinants; Educational Interventions; Primary schools
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children attending primary school: In this study will be included children 6-11 years and their families, whose parents will provide written consent to participate,
  Interventions: Behavioral: Educational interventions

INTERVENTIONS:
Behavioral: Educational interventions — The educational interventions will consist in:

SUMMARY:
Childhood obesity condition has increased 10 times in the last 40 years, representing one of the most important public health challenges of our century.

The overweight and obesity in children are conditions associated with several determinants, mostly related to dietary habits, physical activity, and environmental behavior.

To counteract childhood obesity, several prevention programs have been promoted, however evidence concerning their efficacy was contrasting, especially among the younger population and in the long term.

Moreover, due to the wide variety of interventions administered it is not clear which specific strategy (or combinations of strategies) was the most effective.

The LIVELY study aims 1) to assess the prevalence and the factors associated to childhood overweight and obesity; 2) to develop multidimensional strategies for prevention of childhood obesity by involving families and recognizing the role of schools as an environment for raising awareness on healthy and sustainable dietary patterns and lifestyle.

DETAILED DESCRIPTION:
LIVELY is a study with a one group pre-test - post-test design (without control). The study will be conducted in the primary schools of the Istituto Luigi Cadorna in Milano (Lombardy Region, Northern Italy). The study population will involve children (6-11 years) belonging to different socioeconomic status and ethnic groups, attending classes of the school whose teachers will accept to participate.

The educational interventions will consist in:

ELIGIBILITY:
Inclusion Criteria:

* children 6-11 years
* children whose parents will provide written consent to participate.

Exclusion Criteria:

* Children who do not have inclusion criteria.

Ages: 6 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: The study population will involve children 6-11 years old, attending the primary school Istituto Luigi Cadorna in Milano (Lombardy Region -Northern Italy) and their families.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Investigate prevalence of childhood overweight and/or obesity | Baseline
  Weight and height will be combined to report BMI in kg/m^2
Investigation on adherence to Mediterranian diet | Baseline
  Mediterranean Diet Quality Index for children and adolescents (KIDMED) will be used. The index ranges from 0 to 12 and is based on 16 questions. The sums of the values from the test are classified into three levels: scores ≥8 are considered optimal, 4-7 as average Mediterranean Diet adherence, and ≤3 as very low diet quality.
Assessment of the consumption of ultra-processed food by children | Baseline
  NOVA classification, which will classify ultra-processed foods in four groups according to their level of processing (Group 1: unprocessed foods - Group 4: ultra-processed foods)
Investigation of family lifestyles | Baseline
  Children Feeding Questionnaire (CFQ) will be used. It measures parental feeding practices and attitudes. The CFQ contains originally 31 items and measures the following seven factors: Perceived Responsibility (three items), Parent Perceived Weight (four items), Perceived Child Weight (six items), Parents Concern about Child Weight (three items), Parents' feeding practices: Restriction (eight items), Pressure to Eat (four items), and Monitoring (three items). The responses to all items are coded on a 5-point Likert scale ranging from one to five.

SECONDARY OUTCOMES:
Feasibility of multidimensional school-based educational interventions | 6 months
  Perception of usefulness of the interventions: appreciation questionnaires to investigate the satisfaction of the implemented activities; organization of the interventions and usefulness of the educational interventions
Investigation of changes in adherence to Mediterranian diet | Baseline, 6 and 12 months
  Mediterranean Diet Quality Index for children and adolescents (KIDMED) will be used. The index ranges from 0 to 12 and is based on 16 questions. The sums of the values from the test are classified into three levels: scores ≥8 are considered optimal, 4-7 as average Mediterranean Diet adherence, and ≤3 as very low diet quality.
Assessment of changes of the consumption of ultra-processed food by children | Baseline, 6 and 12 months
  NOVA classification, which will classify ultra-processed foods in four groups according to their level of processing (Group 1: unprocessed foods - Group 4: ultra-processed foods)
Investigation of changes of family lifestyles | Baseline, 6 and 12 months
  Children Feeding Questionnaire (CFQ) will be used. It measures parental feeding practices and attitudes. The CFQ contains originally 31 items and measures the following seven factors: Perceived Responsibility (three items), Parent Perceived Weight (four items), Perceived Child Weight (six items), Parents Concern about Child Weight (three items), Parents' feeding practices: Restriction (eight items), Pressure to Eat (four items), and Monitoring (three items). The responses to all items are coded on a 5-point Likert scale ranging from one to five.

CONTACTS AND LOCATIONS:
Overall Officials: Carlotta Franchi, PhD, Principal Investigator — Mario Negri Institute for Pharmacological Research; Marta Baviera, PharmDr, Principal Investigator — Mario Negri Institute for Pharmacological Research; Maria Vittoria Conti, MSc, Principal Investigator — University of Pavia
Locations (1):
- Istituto Comprensivo Luigi Cadorna, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Basilico S, Conti MV, Ardoino I, Breda C, Loperfido F, Klaic E, Spialtini L, Foresta A, Orsini F, Ojeda Fernandez ML, Conca Bonizzoni S, Modena E, Tootoonchi Hamedani Y, Villa F, Cena H, Baviera M, Franchi C. Multidimensional School-Based and Family-Involved Interventions to Promote a Healthy and Sustainable Lifestyle (LIVELY) for Childhood Obesity Prevention: Study Protocol. JMIR Res Protoc. 2024 Oct 30;13:e57509. doi: 10.2196/57509. PMID 39475855